CLINICAL TRIAL: NCT01130194
Title: A Pilot Phase II Study Of Sequential Treatment With Chemotherapy, Radioimmunotherapy and Autologous Hematopoietic Stem Cell Transplantation in Patients With Follicular Lymphoma
Brief Title: Immunochemotherapy, Zevalin, and Bone Marrow Transplant for Follicular Lymphoma
Acronym: MasterPlan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #14228
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; radioimmunotherapy; rituximab; C-MOPP-R; autologous transplant
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cyclophosphamide; Rituximab; Vincristine; Procarbazine; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): C-MOPP-R chemotherapy, 6 cycles Peripheral blood stem cell mobilization Radioimmunotherapy Autologous Hematopoietic Stem Cell Transplantation
  Interventions: Other: Combination of treatment modalities

INTERVENTIONS:
Other: Combination of treatment modalities — Intravenous cyclophosphamide, rituximab, and vincristine day 1 and 8 of 28 day cycles for 6 cycles total.
  Oral prednisone and procarbazine day 1-14 of every 28 day cycle. Yttrium ibritumomab tiuxetan intravenous injection. Autologous stem cell transplant with intravenous BEAM (BCNU or carmustine, etoposide, ara-C or cytarabine, melphalan) chemotherapy conditioning.
  Other Names: Cytoxan; Rituxan; Oncovin; Matulane; Zevalin

SUMMARY:
Follicular lymphoma has historically been considered an incurable lymphoma. By combining multiple effective treatments, the investigators believe that prolonged disease-free survival is achievable in this disease. The investigators goal is to have at least 60-70% of our patients in first continuous complete remission 15 years from initiation of treatment.

DETAILED DESCRIPTION:
Patients will receive six cycles of combination chemotherapy, C-MOPP-R, typically through a subcutaneous PORT. This combination chemotherapy will last six months. After the last dose of chemotherapy, patients will have a 2 month treatment holiday prior to undergoing stem cell mobilization from peripheral blood with subcutaneous injections of neupogen and mozobil. Patients then receive Zevalin radioimmunotherapy, and this is followed after recovery of blood counts, typically 3 months later, by an autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Follicular lymphoma, newly diagnosed or previously treated but no more than 2 previous regimens
* Relapse of disease must be greater than 6 months after last chemotherapy
* Stages II, III or IV
* Eastern Cooperative Group (ECOG) performance status of 0 or 1. If ECOG 2-4, poor performance must by due to lymphoma as judged by study investigator.
* Patient signed written informed consent
* Adequate renal function defined as a glomerular filtration rate (GFR) > 60 ml/min
* Adequate blood counts (absolute neutrophil count ≥ 1,500, platelets ≥100,000), unless low due to lymphomatous involvement of the bone marrow.
* No known allergies to the chemotherapeutic agents
* No other major disabling co morbidities
* Adequate pulmonary function, defined as corrected DLCO greater than 70% of predicted and FEV1 (forced expiratory volume in one second, a test of respiratory function) greater than 50% of predicted.
* Adequate hepatic function as assessed by study investigator
* Adequate cardiac function, defined as baseline MUGA (Multiple gated acquisition, a test of heart function) >50%

Exclusion Criteria:

* Stage I follicular lymphoma
* ECOG performance status ≥ 2, unless due to lymphoma
* Patient refuses to sign written informed consent
* Poor renal function defined as GFR <60ml/min
* Abnormal liver function as assessed by study investigator
* Poor bone marrow reserve (absolute neutrophil count <1,500 and/or platelets < 100,000) not attributable to lymphomatous involvement of the bone marrow.
* Hypersensitivity to the chemotherapeutic agents
* Major disabling co morbidities like uncontrolled severe HTN (hypertension), active coronary artery disease, liver cirrhosis.
* Previously diagnosed malignancy other than basal or squamous cell carcinoma of the skin diagnosed <5 years prior.
* Central nervous system disease
* History of advanced cardiac disease (Active angina, Congestive heart failure with a LVEF (left ventricular ejection fraction) <50%).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival percentage(intention to treat) | 5 years

SECONDARY OUTCOMES:
Incidence of second malignancies | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Petruska, MD, Principal Investigator — St. Louis University; Mark J Fesler, MD, Study Director — St. Louis University
Locations (1):
- Saint Louis University Cancer Center, St Louis, Missouri, United States

REFERENCES:
- [Result] Fesler MJ, Osman M, Glauber J, Petruska PJ. C-MOPP: Results of a Forgotten Regimen in the Era of Rituximab and PET. Blood (ASH Annual Meeting Abstracts 2009) #4577.